CLINICAL TRIAL: NCT06297681
Title: A Cross-sectional Study on the Efficacy and Safety of the Combination of Daratumumab+Bortezomib+Dexamethasone Regimen and Dapagliflozin in the Treatment of M-protein Related Cardiac Disease
Brief Title: Combination of Daratumumab and BD Regimen and Dapagliflozin in the Treatment of M-protein Related Cardiac Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Chuiyangliu Hospital (Other Government); Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1-27-2
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: M-protein Related Cardiac Disease
Keywords: M-protein related cardiac disease; daratumumab; dapagliflozin; bortezomib; dexamethasone
MeSH Terms: interventions — daratumumab; Bortezomib; Dexamethasone; dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, urine, bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed M-protein related cardiac disease group: M-protein related cardiac disease aged 18 and above (at least one of the following criteria is met): (1) Systemic amyloidosis of the affected heart; (2) Presence of M component and presence of arrhythmia, cardiac enzyme abnormalities, cardiac function abnormalities, and exclusion of other diagnosable cardiac diseases. It is expected to include 40 patients with M-protein related cardiac disease. The treatment medication for enrolled patients must comply with the treatment regimen of Daratumumab + Bortezomib + Dexamethasone. All patients were given Dapagliflozin 10mg/day at the beginning of treatment (creatinine clearance rate greater than 20ml/min).
  Interventions: Drug: Daratumumab + Bortezomib + Dexamethasone + Dapagliflozin

INTERVENTIONS:
Drug: Daratumumab + Bortezomib + Dexamethasone + Dapagliflozin — The treatment medication for enrolled patients must comply with the treatment regimen of Daratumumab + Bortezomib + Dexamethasone: subcutaneous injection of 1800mg of Daratumumab, d1, 8,15,22 (28 day cycle); (After 2 cycles of improvement in cardiac indicators, it can be adjusted to intravenous injection of daratumumab); Bortezomib 1.3 mg/m2 d1, 8, 15, 22; D1, 8, 15, 22; Dexamethasone 20 mg d1, 2, 8, 9, 15, 16, 22, 23. When NTProBNP is greater than 5400ng/ml, bortezomib 1.0mg/m2; When NTProBNP is greater than 8500ng/ml, bortezomib is 0.7mg/m2. When NTProBNP is greater than 10000ng/ml, bortezomib is temporarily not allowed; NTProBNP greater than 4500ng/ml dexamethasone starts at 10 mg/dose. All patients were given Dapagliflozin 10mg/day at the beginning of treatment (creatinine clearance rate greater than 20ml/min).

SUMMARY:
It is expected to include 40 patients with M-protein related cardiac disease. The treatment medication for enrolled patients must comply with the treatment regimen of Daratumumab + Bortezomib + Dexamethasone. All patients were given Dapagliflozin 10mg/day at the beginning of treatment (creatinine clearance rate greater than 20ml/min).

DETAILED DESCRIPTION:
This study is a multicenter, single arm, observational clinical study.It is expected to include 40 patients with M-protein related cardiac disease, who will sign informed consent forms. Collect baseline examination, treatment period (planned 6 cycles), and follow-up period (survival follow-up) data for patients who meet the inclusion and exclusion criteria. The treatment medication for enrolled patients must comply with the treatment regimen of Daratumumab + Bortezomib + Dexamethasone: subcutaneous injection of 1800mg of Daratumumab, d1, 8,15,22 (28 day cycle); (After 2 cycles of improvement in cardiac indicators, it can be adjusted to intravenous injection of daratumumab); Bortezomib 1.3 mg/m2 d1, 8, 15, 22; D1, 8, 15, 22; Dexamethasone 20 mg d1, 2, 8, 9, 15, 16, 22, 23. When NTProBNP is greater than 5400ng/ml, bortezomib 1.0mg/m2; When NTProBNP is greater than 8500ng/ml, bortezomib is 0.7mg/m2. When NTProBNP is greater than 10000ng/ml, bortezomib is temporarily not allowed; NTProBNP greater than 4500ng/ml dexamethasone starts at 10 mg/dose. All patients were given Dapagliflozin 10mg/day at the beginning of treatment (creatinine clearance rate greater than 20ml/min).

ELIGIBILITY:
Inclusion Criteria:

* M-protein related cardiac disease aged 18 and above (at least one of the following criteria is met): (1) Systemic amyloidosis of the affected heart; (2) Presence of M component and presence of arrhythmia, cardiac enzyme abnormalities, cardiac function abnormalities, and exclusion of other diagnosable cardiac diseases;
* ECOG score 0-2;
* Sign a written informed consent form.

Exclusion Criteria:

* Acute myocardial infarction;
* Severe functional abnormalities in important organs such as lungs, liver, and kidneys (the carbon monoxide diffusion ability caused by chronic respiratory diseases is 50% lower than expected);
* Major surgery, radiation therapy, infections requiring systemic antibiotic treatment, or other serious infections within 14 days after enrollment;
* Individuals with mental illness, comprehension disorders, or other reasons that make it difficult to control themselves;
* Pregnant or lactating women, as well as reproductive age patients who refuse to take appropriate contraceptive measures during this trial. If the patient is male, refuse to use adequate contraceptive methods or donate semen during the study period and within 3 months after receiving the last cycle of drug study;
* Diagnosed or treated another malignant tumor within 2 years prior to enrollment;
* Individuals with allergies to daratumumab, bortezomib, or dexamethasone components or more severe allergic constitutions;
* HIV infected individuals (HIV antibody positive);
* Active infection of hepatitis B and hepatitis C (hepatitis B B virus surface antigen positive and/or hepatitis B core antibody positive, hepatitis B virus DNA more than 1x103 copies/mL; hepatitis C virus RNA more than 1x103 copies/mL);
* Participate in another clinical trial 30 days after the start of the trial and throughout the entire trial period;
* The researcher determined that patients who are not suitable to participate in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Observe patient data from Beijing Chaoyang Hospital affiliated with Capital Medical University, Beijing Chuiyangliu Hospital, and Beijing Boren Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | After 6 cycles of treatment (28 days as 1 cycle)
  The percentage of cases that achieved complete response (CR) and partial response (PR) after treatment compared to the total evaluable cases.

SECONDARY OUTCOMES:
2-year PFS rate, progression free survival (PFS) | Treatment for 2 years
  The time interval from enrollment to objective observation of disease progression or death (caused by any reason).
2-year OS rate, overall survival (OS) | Treatment for 2 years
  The time from enrollment to death due to any reason. For non deceased subjects, the cut-off date will be the last known survival date of the subjects.
Duration of Relief (DOR) | Treatment for 2 years
  The time from the first assessment of the tumor as CR or PR to the first assessment as PD (Progressive Disease) or death from any cause.
Next treatment time (TTNT) | Treatment for 2 years
  The time interval from enrollment to receiving subsequent treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kastritis E, Palladini G, Minnema MC, Wechalekar AD, Jaccard A, Lee HC, Sanchorawala V, Gibbs S, Mollee P, Venner CP, Lu J, Schonland S, Gatt ME, Suzuki K, Kim K, Cibeira MT, Beksac M, Libby E, Valent J, Hungria V, Wong SW, Rosenzweig M, Bumma N, Huart A, Dimopoulos MA, Bhutani D, Waxman AJ, Goodman SA, Zonder JA, Lam S, Song K, Hansen T, Manier S, Roeloffzen W, Jamroziak K, Kwok F, Shimazaki C, Kim JS, Crusoe E, Ahmadi T, Tran N, Qin X, Vasey SY, Tromp B, Schecter JM, Weiss BM, Zhuang SH, Vermeulen J, Merlini G, Comenzo RL; ANDROMEDA Trial Investigators. Daratumumab-Based Treatment for Immunoglobulin Light-Chain Amyloidosis. N Engl J Med. 2021 Jul 1;385(1):46-58. doi: 10.1056/NEJMoa2028631. PMID 34192431
- [Background] Suzuki K, Wechalekar AD, Kim K, Shimazaki C, Kim JS, Ikezoe T, Min CK, Zhou F, Cai Z, Chen X, Iida S, Katoh N, Fujisaki T, Shin HJ, Tran N, Qin X, Vasey SY, Tromp B, Weiss BM, Comenzo RL, Kastritis E, Lu J. Daratumumab plus bortezomib, cyclophosphamide, and dexamethasone in Asian patients with newly diagnosed AL amyloidosis: subgroup analysis of ANDROMEDA. Ann Hematol. 2023 Apr;102(4):863-876. doi: 10.1007/s00277-023-05090-z. Epub 2023 Mar 2. PMID 36862168
- [Background] Minnema MC, Dispenzieri A, Merlini G, Comenzo RL, Kastritis E, Wechalekar AD, Grogan M, Witteles R, Ruberg FL, Maurer MS, Tran N, Qin X, Vasey SY, Weiss BM, Vermeulen J, Jaccard A. Outcomes by Cardiac Stage in Patients With Newly Diagnosed AL Amyloidosis: Phase 3 ANDROMEDA Trial. JACC CardioOncol. 2022 Nov 15;4(4):474-487. doi: 10.1016/j.jaccao.2022.08.011. eCollection 2022 Nov. PMID 36444227
- [Background] Sanchorawala V, Palladini G, Minnema MC, Jaccard A, Lee HC, Gibbs S, Mollee P, Venner C, Lu J, Schonland S, Gatt M, Suzuki K, Kim K, Cibeira MT, Beksac M, Libby E, Valent J, Hungria V, Wong SW, Rosenzweig M, Bumma N, Chauveau D, Gries KS, Fastenau J, Tran NP, Qin X, Vasey SY, Weiss BM, Vermeulen J, Ho KF, Merlini G, Comenzo RL, Kastritis E, Wechalekar AD. Health-related quality of life in patients with light chain amyloidosis treated with bortezomib, cyclophosphamide, and dexamethasone +/- daratumumab: Results from the ANDROMEDA study. Am J Hematol. 2022 Jun 1;97(6):719-730. doi: 10.1002/ajh.26536. Epub 2022 Mar 30. PMID 35293006
- [Background] Wechalekar AD, Cibeira MT, Gibbs SD, Jaccard A, Kumar S, Merlini G, Palladini G, Sanchorawala V, Schonland S, Venner C, Boccadoro M, Kastritis E. Guidelines for non-transplant chemotherapy for treatment of systemic AL amyloidosis: EHA-ISA working group. Amyloid. 2023 Mar;30(1):3-17. doi: 10.1080/13506129.2022.2093635. Epub 2022 Jul 15. PMID 35838162